CLINICAL TRIAL: NCT01252654
Title: Comparison of Intralase and Visumax Femtosecond Laser for Laser In Situ Keratomileusis
Status: Completed | Type: Observational
Sponsor: Singapore Eye Research Institute (Other)
Responsible Party: Principal Investigator, Jodhbir Mehta, Head Tissue Engineering and Stem Cell Group, Singapore Eye Research Institute
Other Study IDs: R683/33/2009; Other (Other Grant/Funding Number: [NMRC/TCR/002 - SERI/2008 - TCR 621/41/2008])
Record Dates: First submitted 2010-05-10; First posted 2010-12-03 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Myopia
Keywords: Lasik; Femtosecond Laser; Visumax; IntraLase; Myopia; Myopic Patients undergoing LASIK
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1 IntraLase flaps: Patients who have undergone flap creation with IntraLase laser
- 2 Visumax flaps: Patients who have undergone flaps created with Visumax laser

SUMMARY:
Emtosecond lasers are used in cutting the flap in LASIK procedures (laser corrective surgery for refractive error). Their use has decreased the incidence of serious complications when compared to the use of microkeratomes(mechanical blades). The commonest femtosecond laser currently used is 'Intralase'. A newer femtosecond laser 'Visumax' (Zeiss) is now available and differs from the Intralase in that it does not interfere with the curvature of the cornea when creating the flap. The Intralase applanates the cornea flat during flap creation which causes the intraocular pressure to be higher. Both Intralase and Visumax lasers are available to patients and surgeons to use at SNEC. The aim of the investigators study is to compare the two lasers in a randomization of left and right eyes in the same patient. The investigators want to measure any difference that the lower intraocular pressure may have during the creation of the flap. This will be measured with a questionaire on patient experience during the procedure and the outcomes of vision, refraction, contrast sensitivity, wave-front analysis, tear function,corneal sensation and flap thickness measured with anterior segment OCT during the post-operative follow up period. To date no-one has compared the use of these two femtosecond lasers. Both lasers are currently used clinically for flap creation at SNEC.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older.
* Cycloplegic spherical equivalent of >-1.00D
* Refractive cylinder -4.00 D or less.
* Best spectacle corrected visual acuity (BSCVA) of 6/12 or better in BOTH eyes.
* Spherical or cylindrical error has progressed at -0.50D or less per year from date of baseline measurement.
* Contact lens wearers must have removed contact lenses at least two (2) weeks before the baseline measurement.
* No evidence of irregular astigmatism on corneal topography.
* Available to attend post-operative examinations for a 3 month period.

Exclusion Criteria:

* Progressive or unstable myopia and/or astigmatism.
* Clinical or corneal topographic evidence of keratoconus.
* Residual, recurrent or active ocular disease such as uveitis, severe dry eyes, severe allergic eye disease, glaucoma, visually significant cataract and retinal disease.
* Previous corneal surgery or trauma within the corneal flap zone.
* Patent corneal vascularization within 1mm of the corneal flap zone.
* Taking systemic medications likely to affect wound healing, such as corticosteroids and antimetabolites.
* Systemically immunocompromised.
* Systemic disease likely to affect wound healing, such as diabetes, connective tissue disease and severe atopy.
* Pregnant or nursing.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Myopic patients presenting to refractive service eligible for LASIK
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2010-01; Primary Completion 2012-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 3 months

SECONDARY OUTCOMES:
complications | 3 months
Subjective questionnaire | 1 weekd
Corneal Sensation | 3 months
Tear function | 3 months
Wavefront analysis | 3 months
Contrast Sensitivity | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Donald Tan, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore

REFERENCES:
- [Derived] D'Souza S, Petznick A, Tong L, Hall RC, Rosman M, Chan C, Koh SK, Beuerman RW, Zhou L, Mehta JS. Comparative analysis of two femtosecond LASIK platforms using iTRAQ quantitative proteomics. Invest Ophthalmol Vis Sci. 2014 May 6;55(6):3396-402. doi: 10.1167/iovs.14-14113. PMID 24801511